CLINICAL TRIAL: NCT04225117
Title: An Open-label, Multicenter, Multicohort, Phase 2 Study to Evaluate Enfortumab Vedotin in Subjects With Locally Advanced or Metastatic Malignant Solid Tumors (EV-202)
Brief Title: A Study to Evaluate Enfortumab Vedotin in Subjects With Locally Advanced or Metastatic Malignant Solid Tumors (EV-202)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Seagen Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7465-CL-202; KEYNOTE-F21 (Other: Merck Sharp & Dohme, LLC); MK-3475-F21 (Other: Merck Sharp & Dohme, LLC); jRCT2080225095 (Registry Identifier: jRCT)
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Locally Advanced or Metastatic Malignant Solid Tumors
Keywords: Squamous NSCLC; Triple negative breast cancer (TNBC); ASG-22CE; non-small cell lung cancer (NSCLC); Hormone receptor-positive/ human epidermal growth factor receptor 2-negative (HR+/HER2-) breast cancer; non-squamous NSCLC; locally advanced or metastatic malignant solid tumors; Head and neck cancer; EV-202; Gastric or gastroesophageal junction (GEJ) or esophageal cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Head and Neck Neoplasms; Esophageal Neoplasms | interventions — enfortumab vedotin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1: HR+/HER2- breast cancer (Experimental): Participants will receive enfortumab vedotin as an intravenous (IV) infusion on days 1, 8 and 15 of each 28-day cycle.
  HR+/HER2- = Hormone receptor-positive/ human epidermal growth factor receptor 2-negative
  Interventions: Drug: enfortumab vedotin
- Cohort 2: Triple negative breast cancer (TNBC) (Experimental): Participants will receive enfortumab vedotin as an intravenous (IV) infusion on days 1, 8 and 15 of each 28-day cycle.
  Interventions: Drug: enfortumab vedotin
- Cohort 3: Squamous non-small cell lung cancer (Experimental): Participants will receive enfortumab vedotin as an intravenous (IV) infusion on days 1, 8 and 15 of each 28-day cycle.
  Interventions: Drug: enfortumab vedotin
- Cohort 4: Non-squamous non-small cell lung cancer (Experimental): Participants will receive enfortumab vedotin as an intravenous (IV) infusion on days 1, 8 and 15 of each 28-day cycle.
  Interventions: Drug: enfortumab vedotin
- Cohort 5: Head and neck cancer (Experimental): Participants will receive enfortumab vedotin as an intravenous (IV) infusion on days 1, 8 and 15 of each 28-day cycle.
  Interventions: Drug: enfortumab vedotin
- Cohort 6: Gastric or GEJ or esophageal cancer (Experimental): Participants enrolled into Cohort 6 will be reallocated based on disease type and histology into Cohorts 7 or 8.
  GEJ= gastroesophageal junction
  Interventions: Drug: enfortumab vedotin
- Cohort 7: Gastric and esophageal adenocarcinoma (EAC) including GEJ adenocarcinoma (Experimental): Participants will receive enfortumab vedotin as an intravenous (IV) infusion on days 1, 8 and 15 of each 28-day cycle.
  Interventions: Drug: enfortumab vedotin
- Cohort 8: Esophageal squamous cell carcinoma (ESCC) (Experimental): Participants will receive enfortumab vedotin as an intravenous (IV) infusion on days 1, 8 and 15 of each 28-day cycle.
  Interventions: Drug: enfortumab vedotin
- Cohort 9: Head and neck squamous cell carcinoma (HNSCC) (Experimental): Participants will receive enfortumab vedotin as an IV infusion on days 1 and 8 of each 21-day cycle. Pembrolizumab will be administered as an IV infusion on day 1 of each 21-day cycle.
  Interventions: Drug: enfortumab vedotin; Drug: pembrolizumab

INTERVENTIONS:
Drug: enfortumab vedotin — intravenous (IV) infusion
  Other Names: ASG-22CE
Drug: pembrolizumab — IV infusion
  Other Names: KEYTRUDA®
  Arms: Cohort 9: Head and neck squamous cell carcinoma (HNSCC)

SUMMARY:
The primary purpose of this study is to determine the antitumor activity of enfortumab vedotin as measured by confirmed objective response rate (ORR) per RECIST v1.1.

This study will also assess other measures of antitumor activity; overall survival (OS); as well as the safety and tolerability of enfortumab vedotin for cohorts 1 to 8 and enfortumab vedotin + pembrolizumab in cohort 9.

DETAILED DESCRIPTION:
This study will consist of 3 periods: screening/baseline, treatment and follow-up.

Screening/baseline period will take place up to 28 days prior to the first dose of study treatment.

In the treatment period, starting at cycle 1, participants in cohorts 1 to 8 will receive enfortumab vedotin on days 1, 8, and 15 every 28-day cycle until one of the treatment discontinuation criteria are met. participants in cohort 9 will receive enfortumab vedotin on days 1, 8, and pembrolizumab on day 1 of every 21-day cycle until one of the treatment discontinuation criteria are met. Disease assessment will be performed at screening/baseline and repeated every 8 weeks (56 days ± 7 days) for cohorts 1 to 8 and first assessment at week 9 and thereafter every 6 weeks (42 days ± 7 days) for cohort 9 from the first dose of study treatment throughout the study until the participant has radiologically confirmed disease progression, initiates a new subsequent anticancer therapy, dies, withdraws consent, is lost to follow-up or the study closes, whichever occurs first.

Participants who discontinue study treatment for reasons other than radiologically-confirmed disease progression by RECIST Version 1.1 will enter into a post treatment follow-up period and continue to receive imaging scans every 8 weeks (56 days ± 7 days) for cohorts 1 to 8 and for cohort 9 first scan will be performed at 9 week and thereafter every 6 weeks (42 days ± 7 days) until the subject has radiologically confirmed disease progression (for cohort 9 confirmed progressive disease [iCPD] per modified RECIST 1.1 for immune-based therapeutics [iRECIST]), initiates a new anticancer therapy, dies, withdraws consent, is lost to follow-up or the study closes, whichever occurs first.

After 1 year on study treatment, the frequency of disease assessment will be reduced to every 12 weeks (84 days ± 7 days) for cohorts 1 to 8.

After 18 months on study treatment, the frequency of disease assessment will be reduced to every 9 weeks (63 days ± 7 days) for cohort 9.

Participants in cohorts 1to 8 who discontinue study treatment for reasons other than radiologically-confirmed disease progression by RECIST Version 1.1 will enter into a post treatment follow-up period and continue to receive imaging scans every 8 weeks (56 days ± 7 days).

Participants in cohort 9 who discontinue study treatment for reasons other than radiologically confirmed disease progression per iRECIST will enter into a post treatment follow-up period and have physical exams, ECOG and disease assessments every 6 weeks (± 7 days) up to 18 months after first dose, then every 9 weeks (± 7 days) until the subject has radiologically confirmed disease progression per iRECIST.

After radiologically-confirmed disease progression or initiation of subsequent anticancer therapy, whichever occurs first, participants will be contacted every 12 weeks in the long-term follow-up period for survival status until death, withdrawal of consent, lost to follow-up or study closure, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Subject is considered an adult according to local regulation at the time of signing the informed consent form (ICF).
* Subject has measurable disease by RECIST Version 1.1.
* Subject has accessible archival tumor tissue from either the primary tumor or a metastatic site, for which source and availability have been confirmed prior to study treatment. If no archival tumor tissue is available, the subject will have a biopsy to obtain tumor tissue prior to study treatment. If the subject is unable to undergo a biopsy due to safety concerns, enrollment into the study must be discussed with the medical monitor.
* For cohort 9 only: Subject should submit archival or fresh tumor tissue sample for programmed cell death-ligand 1 (PD-L1) central testing during screening if no local PD-L1 test result is available. Central test result for PD-L1 will be required prior to subject enrollment. For cohort 9 subjects with local PD-L1 test result confirming CPS ≥ 1, archival or fresh tissue sample for exploratory analysis should be submitted within 5 days of enrollment.
* Subject has ECOG performance status of 0 or 1.
* Subject has the following baseline laboratory data. If a subject has received a recent blood transfusion, the hematology tests must be obtained ≥ 28 days after any blood transfusion.

  * absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L
  * platelet count ≥ 100 × 10^9/L
  * hemoglobin ≥ 9 g/dL
  * serum total bilirubin ≤ 1.5 × upper limit of normal (ULN) or ≤ 3 × ULN for subjects with Gilbert's disease
  * creatinine clearance (CrCl) ≥ 30 mL/min as estimated per institutional standards or as measured by 24-hour urine collection (glomerular filtration rate [GFR] can also be used instead of CrCl).
  * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN
* Subject agrees not to participate in another interventional study while receiving study treatment in the present study.
* Additional contraceptive requirements exist for male and female subjects.

Disease Specific Inclusion Criteria:

* Evidence of progression on or after the last regimen received.
* Locally advanced or metastatic disease that is not amenable to curative intent treatment.

Cohort 1: HR+/HER2- breast cancer

* Subject has evidence of radiographic progression on or after the last regimen received.
* Subject has histologically- or cytologically-confirmed HR+/HER2- (estrogen receptor [ER] positive and/or progesterone receptor [PR] positive, and HER2 negative) breast cancers and are not considered a candidate for further hormonal therapy. Subject will be considered HR+ if biopsies show ≥ 1% expression of ER or PR as per current American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines.
* Subject has locally advanced or metastatic disease that is not amenable to curative intent treatment.
* Subject must have received a taxane or anthracycline in the neoadjuvant, adjuvant or incurable, locally advanced or metastatic setting.

  * Prior cytotoxic regimen received in the neoadjuvant or adjuvant setting will count as a prior cytotoxic regimen if disease recurrence occurred during or within 6 months of completing the regimen.
* Subject has progressed, relapsed, or discontinued for toxicity during or after at least 1 prior standard of care cytotoxic regimen in the incurable, unresectable locally advanced or metastatic setting, and has not received > 2 prior lines of cytotoxic therapy in the locally advanced or metastatic setting. No limit applies to endocrine therapies. Poly(ADP-ribose) polymerases (PARP) inhibitors do not count as a line of cytotoxic therapy.
* Subject has progressed, relapsed, or discontinued for toxicity during or after receiving endocrine therapy or with hormonally-directed therapy with cyclin-dependent kinase (CDK) inhibitors. Prior therapy with CDK inhibitors is not required.

Cohort 2: triple negative breast cancer (TNBC)

* Subject has evidence of radiographic progression on or after the last regimen received.
* Subject has histologically- or cytologically-confirmed TNBC; defined as unequivocal TNBC histology (ER-negative/PR-negative/HER2-negative). This is defined by < 1% expression of ER and PR by immunohistochemistry (IHC), and that are, for HER2, either 0 to 1+ by IHC, or IHC 2+ and fluorescence in situ hybridization (FISH) negative (not amplified) as per current ASCO/CAP guidelines.
* Subject has locally advanced or metastatic disease that is not amenable to curative intent treatment.
* Subject must have received a taxane or anthracycline in the neoadjuvant, adjuvant or incurable, locally advanced or metastatic setting.

  * Prior cytotoxic regimen received in the neoadjuvant or adjuvant setting will count as a prior cytotoxic regimen if disease recurrence occurred during or within 6 months of completing the regimen.
* Subject has progressed, relapsed, or discontinued for toxicity during or after at least 1 prior standard of care cytotoxic regimen in the incurable, unresectable locally advanced or metastatic setting, and has not received > 2 prior lines of cytotoxic therapy in the locally advanced or metastatic setting. Poly(ADP-ribose) polymerases (PARP) inhibitors do not count as a line of cytotoxic therapy.
* Subject has received prior therapy with an anti-programmed cell death protein-1 (PD-1) or an anti-programmed cell death-ligand 1 (PD-L1) based on subject's tumor PD-1 or PD-L1 expression and local treatment guidelines and has progressed or discontinued treatment due to toxicity, or therapy is contraindicated for subject.

Cohort 3: squamous non-small cell lung cancer (NSCLC)

* Subject has evidence of radiographic progression on or after the last regimen received.
* Subject has histologically or cytologically-confirmed squamous NSCLC.

  * Subjects with mixed histology NSCLC are eligible provided there is not any component of neuroendocrine histology.
  * Subjects with known epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), reactive oxygen species (ROS), BRAF, or other actionable mutations are eligible if treated with mutation targeted therapy and have progressed, relapsed, or discontinued treatment due to toxicity.
* Subject has locally advanced or metastatic disease that is not amenable to curative intent treatment.
* Subject has progressed, relapsed, or discontinued treatment due to toxicity after 1 platinum-based standard of care regimen for locally advanced or metastatic disease, and has not received > 2 prior lines of cytotoxic anticancer therapy in the locally advanced or metastatic setting.

  1. Subjects with locally advanced disease who previously received curative intent treatment with platinum-based standard of care regimen in the adjuvant or neoadjuvant setting or as part of concomitant chemoradiation therapy are eligible if they have progressed or relapsed within 6 months of completion.
  2. Maintenance therapy does not constitute a new chemotherapy regimen provided there was no progression after the initial platinum-based regimen.
  3. Changing chemotherapy agents during platinum-based treatment for the management of toxicities does not constitute a new chemotherapy regimen provided no progression had occurred while on the initial therapy.
* Subject has received prior therapy with an anti-PD-1 or anti-PD-L1 based on subject's tumor PD-1 or PD-L1 expression and local treatment guidelines and has progressed, relapsed, or discontinued treatment due to toxicity, or therapy is contraindicated for subject.

Cohort 4: non-squamous non-small cell lung cancer

* Subject has evidence of radiographic progression on or after the last regimen received.
* Subject has histologically- or cytologically-confirmed non-squamous NSCLC.

  * Subjects with mixed histology NSCLC are eligible provided there is not any component of neuroendocrine histology.
  * Subjects with known EGFR, ALK, ROS, BRAF, or other actionable mutations are eligible if treated with mutation targeted therapy and have progressed, relapsed, or discontinued treatment due to toxicity.
* Subject has locally advanced or metastatic disease that is not amenable to curative intent treatment.
* Subject has progressed, relapsed, or discontinued treatment due to toxicity after 1 platinum-based standard of care regimen for locally advanced or metastatic disease, and has not received > 2 prior lines of cytotoxic anticancer therapy in the locally advanced or metastatic setting.

  1. Subjects with locally advanced disease who previously received curative intent treatment with platinum-based standard of care regimen in the adjuvant or neoadjuvant setting or as part of concomitant chemoradiation therapy are eligible if they have progressed or relapsed within 6 months of completion.
  2. Maintenance therapy does not constitute a new chemotherapy regimen provided there was no progression after the initial platinum-based regimen.
  3. Changing chemotherapy agents during platinum-based treatment for the management of toxicities does not constitute a new chemotherapy regimen provided no progression has occurred while on the initial therapy.
* Subject has received prior therapy with an anti-PD-1 or anti-PD-L1 based on subject's tumor PD-1 or PD-L1 expression and local treatment guidelines and has progressed, relapsed, or discontinued treatment due to toxicity, or therapy is contraindicated for subject.

Cohort 5: second-line or later head and neck cancer

* Subject has evidence of radiographic progression on or after the last regimen received.
* Subject has histologically- or cytologically-confirmed head and neck cancer.

  * Primary tumor site must arise from the oral cavity, oropharynx, hypopharynx, and larynx; tumors arising from the nasopharynx are excluded. Salivary gland tumors and/or parotid gland tumors are not eligible for Cohort 5.
* Subject has locally advanced or metastatic disease that is not amenable to curative intent treatment.
* Subject has progressed, relapsed, or discontinued treatment due to toxicity after 1 platinum-based standard of care regimen for locally advanced or metastatic disease, and has not received > 2 prior lines of cytotoxic anticancer therapy in the locally advanced or metastatic setting.

  * Subjects with locally advanced disease who previously received curative intent treatment with platinum-based standard of care regimen in the adjuvant or neoadjuvant setting or as part of concomitant chemoradiation therapy are eligible if they have progressed or relapsed within 6 months after completion.
* Subject has received prior therapy with an anti-PD-1 or anti-PD-L1 based on subject's tumor PD-1 or PD-L1 expression and local treatment guidelines and has progressed, relapsed, or discontinued treatment due to toxicity, or therapy is contraindicated for subject.

Cohorts 6, 7 and 8: gastric or gastroesophageal junction (GEJ) or esophageal adenocarcinoma

* Subject has evidence of radiographic progression on or after the last regimen received.
* Subject has histologically- or cytologically-confirmed gastric, GEJ, or esophageal cancer.
* Subject has locally advanced or metastatic disease that is not amenable to curative intent treatment.
* Subject has progressed, relapsed, or discontinued due to toxicity after 1 platinum-based standard of care regimen for locally advanced or metastatic disease, and has not received > 2 prior lines of cytotoxic anticancer therapy in the locally advanced or metastatic setting.

  * Neoadjuvant or adjuvant cytotoxic regimens will count as a prior regimen if relapsed or progressed ≤ 6 months after completion.
* Subject must have received a HER2 directed therapy if known to have HER2 positive cancer.
* Subject has received prior therapy with an anti-PD-1 or anti-PD-L1 based on subject's tumor PD-1 or PD-L1 expression and local treatment guidelines and has progressed, relapsed, or discontinued treatment due to toxicity, or therapy is contraindicated for subject.

Cohort 9: 1L HNSCC

* Subject has histologically- or cytologically-confirmed head and neck squamous cell carcinoma.

  a. Primary tumor site must arise from the oral cavity, oropharynx, hypopharynx, and larynx; tumors arising from the nasopharynx are excluded. Salivary gland tumors and/or parotid gland tumors are not eligible for Cohort 9.
* Subject has recurrent or metastatic disease that is incurable by local therapies.
* Subject's tumor sample has PD-L1 combined positive score (CPS) of ≥ 1 as determined by local or central IHC testing.
* Subject has had no prior systemic therapy administered with the exception of systemic therapy completed > 6 months prior if given as part of multimodal treatment for locally advanced disease. Subjects who have received a PD-1 or PD-L1 inhibitor in the curative setting are eligible if it has been at least 12 months since last dose of the anti PD-L1 agent.
* Subject has ANC ≥ 1.5 × 10^9/L.
* International normalized ratio (INR) OR prothrombin time (PT) and activated partial thromboplastin (aPTT) both ≤ 1.5 × ULN unless subject is receiving anticoagulant therapy as long as PT or aPTT is within the therapeutic range of intended use of anticoagulants. PTT may be used if local lab is unable to perform aPTT.
* For subjects with oropharynx tumors, subject has results from testing of HPV status by p16 testing.

Exclusion Criteria:

For All Cohorts:

* Subject has preexisting sensory or motor neuropathy Grade ≥ 2.
* Subject has active central nervous system (CNS) metastases. Subjects with treated CNS metastases are permitted on study if all the following are true:

  * CNS metastases have been clinically stable for ≥ 6 weeks prior to screening
  * If requiring steroid treatment for CNS metastases, the subject is on a stable dose ≤ 20 mg/day of prednisone or equivalent for ≥ 2 weeks
  * Baseline imaging scans show no evidence of new or enlarged brain metastasis
  * Subject does not have leptomeningeal disease
* Subject has ongoing clinically significant toxicity (Grade 2 or higher with the exception of alopecia) associated with prior treatment (including systemic therapy, radiotherapy or surgery).
* Subjects with ongoing ≥ Grade 3 immunotherapy-related hypothyroidism or panhypopituitarism are excluded. Subjects with ongoing immunotherapy-related colitis, uveitis, myocarditis or pneumonitis, or subjects with other immunotherapy-related AEs requiring high doses of steroids (> 20 mg/day of prednisone or equivalent), are excluded. Subject with ≤ Grade 2 immunotherapy-related hypothyroidism or panhypopituitarism may be enrolled when well maintained/controlled on a stable dose of hormone replacement therapy (if indicated).
* Subject has a history of uncontrolled diabetes mellitus within 3 months before the first dose of study treatment. Uncontrolled diabetes (within 3 months before first dose) is defined as hemoglobin A1c (HbA1c) ≥ 8% or HbA1c between 7 and < 8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained. The lowest HbA1c during the screening period will be used to determine eligibility.
* Subject has prior treatment with enfortumab vedotin or other monomethyl auristatin E (MMAE) based antibody-drug conjugates (ADCs).
* Subject has a second malignancy diagnosed within 3 years before first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Subjects with non-melanoma skin cancer, localized prostate cancer treated with curative intent with no evidence of progression, low-risk or very low-risk (per standard guidelines) localized prostate cancer under active surveillance/watchful waiting without intent to treat, or carcinoma in situ of any type (if complete resection was performed) are allowed.
* Subject is currently receiving systemic antimicrobial treatment for viral, bacterial, or fungal infection at the time of first dose of study treatment. Routine antimicrobial prophylaxis is permitted.
* Subject has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or active hepatitis C (e.g., hepatitis C virus [HCV] RNA [qualitative] is detected).
* Subject has known history of human immunodeficiency virus (HIV) infection (HIV 1 or 2).
* Subject has documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction or cardiac symptoms (including congestive heart failure) consistent with New York Heart Association Class III-IV within 6 months prior to the first dose of study drug.
* Subject has major surgery within 4 weeks prior to first dose of study drug.
* Subject had radiotherapy, chemotherapy, biologics, investigational agents, and/or antitumor treatment with immunotherapy that is not completed 2 weeks prior to first dose of study drug.
* Subject has known hypersensitivity to enfortumab vedotin or to any excipient contained in the drug formulation of enfortumab vedotin (including histidine, trehalose dihydrate and polysorbate 20) OR subject has known hypersensitivity to biopharmaceutical produced in Chinese hamster ovary cells.
* Subject has known active keratitis or corneal ulcerations. Subject with superficial punctate keratitis is allowed if the disorder is being adequately treated.
* Subject has any condition which makes the subject unsuitable for study participation.

Cohort 9: 1L HNSCC

* Had PD within 6 months of completion of curatively intended systemic treatment for locoregionally advanced HNSCC.
* Has had an allogeneic tissue/solid organ transplant. Has severe hypersensitivity (≥grade 3) to pembrolizumab and/or any of its excipients.
* Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease.
* Has a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Has a life expectancy of less than 3 months and/or has rapidly progressing disease (e.g. tumor bleeding, uncontrolled tumor pain) in the opinion of the treating investigator.
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

  1. Replacement therapy (e.g., thyroxine, insulin, physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
  2. Brief (<7 days) use of systemic corticosteroids is allowed when use is considered standard of care.
  3. Subjects with vitiligo, psoriasis, type 1 diabetes mellitus, hypothyroidism, or resolved childhood asthma/atopy will not be excluded.
  4. Subjects requiring intermittent use of bronchodilators, inhaled steroids, or local steroid injections will not be excluded.
  5. Subjects with hypothyroidism that is stable with hormone replacement or Sjögren's syndrome will not be excluded.
* Has an active infection requiring systemic therapy.
* Has received prior therapy with an anti-PD-1 or anti-PD-L1 agent in the recurrent/metastatic setting. If anti-PD-1 or anti-PD-L1 agent was given as part of curative intent therapy, it must be at least 1 year since last dose.
* Has received a live vaccine within 30 days of planned start of study therapy. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
* Subject has active tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Cohorts 1-8: Confirmed Overall Response Rate (ORR) (Complete Response (CR) and Partial Response(PR)) per RECIST V1.1 per investigator assessment | Up to 3 years
  Confirmed ORR is defined as the proportion of participants whose objective response is a confirmed CR or PR according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 per investigator assessment.
Cohort 9: Confirmed Overall Response Rate (ORR) (Complete Response (CR) and Partial Response (PR)) per RECIST V1.1 per investigator assessment | Up to 3 years
  Confirmed ORR is defined as the proportion of participants whose objective response is a confirmed CR or PR according to RECIST Version 1.1 per investigator assessment.

SECONDARY OUTCOMES:
Cohorts 1-8: Duration of Response (DOR) per RECIST V1.1 as per investigator assessment | Up to 3 years
  DOR is defined as the time from the date of first documented response (CR or PR that is subsequently confirmed) to the date of first documented progressive disease (PD) per RECIST version 1.1 or death due to any cause, whichever occurs first. DOR will only be calculated for participants achieving a confirmed CR or PR.
Cohorts 1-8: Disease Control Rate (DCR) per RECIST V1.1 as per investigator assessment | Up to 3 years
  DCR is defined as the proportion of participants whose Best Overall Response (BOR) is confirmed CR or PR or stable disease (SD).
Cohorts 1-8: Duration of Progression Free Survival (PFS) per RECIST V1.1 as per investigator assessment | Up to 3 years
  PFS is defined as the time from start of study treatment to first documentation of PD per RECIST version 1.1 or death due to any cause, whichever comes first.
Cohorts 1-8: Duration of Overall Survival (OS) | Up to 3 years
  OS is defined as the time from start of study treatment to date of death due to any cause.
Cohorts 1-8: Number of participants with Adverse Events (AEs) | Up to 2 years
  AEs will be coded using medical dictionary for regulatory activities (MedDRA). An AE is any untoward medical occurrence in a participant administered enfortumab vedotin, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of enfortumab vedotin whether or not considered related to the enfortumab vedotin. An AE is considered "serious" if the event: results in death; is life-threatening; results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions; results in congenital anomaly or birth defect; requires inpatient hospitalization (except for planned procedures) or leads to prolongation of hospitalization (except if prolongation of planned hospitalization is not caused by an AE); or other medically important events.
Cohorts 1-8: Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to 2 years
  Number of participants with potentially clinically significant laboratory values.
Cohorts 1-8: Number of participants with vital sign abnormalities and /or adverse events (AEs) | Up to 2 years
  Number of participants with potentially clinically significant vital sign values.
Cohorts 1-8: Number of participants with routine 12-lead electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | Up to 2 years
  Number of participants with potentially clinically significant ECG values.
Cohorts 1-8: Number of participants at each grade of the Eastern Cooperative Oncology Group Performance Status (ECOG PS) | Up to 2 years
  The ECOG scale will be used to assess performance status. Grades range from 0 (equals fully active, able to carry on all pre-disease performance without restriction), and 5 (equals dead).
Cohort 9: Duration of Response (DOR) per RECIST V1.1 as per investigator assessment | Up to 3 years
  DOR is defined as the time from the date of first documented response (CR or PR that is subsequently confirmed) to the date of first documented progressive disease (PD) per RECIST version 1.1 or death due to any cause, whichever occurs first. DOR will only be calculated for participants achieving a confirmed CR or PR.
Cohort 9: Disease Control Rate (DCR) per RECIST V1.1 as per investigator assessment | Up to 3 years
  DCR is defined as the proportion of participants whose Best Overall Response (BOR) is confirmed CR or PR or stable disease (SD).
Cohort 9: Duration of Progression Free Survival (PFS) per RECIST V1.1 as per investigator assessment | Up to 3 years
  PFS is defined as the time from start of study treatment to first documentation of PD per RECIST version 1.1 or death due to any cause, whichever comes first.
Cohort 9: Duration of Overall Survival (OS) | Up to 3.5 years
  OS is defined as the time from start of study treatment to date of death due to any cause.
Cohort 9: Number of participants with Adverse Events (AEs) | Up to 2 years
  AEs will be coded using medical dictionary for regulatory activities (MedDRA). An AE is any untoward medical occurrence in a participant administered enfortumab vedotin, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of enfortumab vedotin whether or not considered related to the enfortumab vedotin. An AE is considered "serious" if the event: results in death; is life-threatening; results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions; results in congenital anomaly or birth defect; requires inpatient hospitalization (except for planned procedures) or leads to prolongation of hospitalization (except if prolongation of planned hospitalization is not caused by an AE); or other medically important events.
Cohort 9: Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to 2 years
  Number of participants with potentially clinically significant laboratory values.
Cohort 9: Number of participants with vital sign abnormalities and /or adverse events (AEs) | Up to 2 years
  Number of participants with potentially clinically significant vital sign values.
Cohort 9: Number of participants with routine 12-lead electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | Up to 2 years
  Number of participants with potentially clinically significant ECG values.
Cohort 9: Number of participants at each grade of the Eastern Cooperative Oncology Group Performance Status (ECOG PS) | Up to 2 years
  The ECOG scale will be used to assess performance status. Grades range from 0 (equals fully active, able to carry on all pre-disease performance without restriction), and 5 (equals dead).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (39):
- United States (29):
  - Arizona Oncology, Tucson, Arizona
  - University of California - San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, Tallahassee, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwestern University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Kansas, Fairway, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - New York University Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Research Center, Dallas, Texas
  - University of Texas, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Site CA15003, Ottawa, Ontario, Canada
- Japan (9):
  - Site JP81004, Nagoya, Aichi-ken
  - Site JP81001, Kashiwa, Chiba
  - Site JP81005, Chuo-ku, Osaka
  - Site JP81007, Ōsaka-sayama, Osaka
  - Site JP81011, Kitaadachi-Gun, Saitama
  - Site JP81006, Nakatogari, Shizuoka
  - Site JP81003, Chūō, Tokyo
  - Site JP81002, Koto, Tokyo
  - Site JP81010, Okayama

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Muro K, Chin K, Maron SB, Braiteh FS, Mitani S, Hara H, Kuboki Y, Mulcahy MF, Baranda JC, Gardner FP, Jin N, Hamauchi S, Kaplan J, Gorla S, Liu S, Wozniak M, Poondru S, Dillon R, Meng C, Kondo S. Phase II trial of enfortumab vedotin in patients with previously treated gastric and esophageal cancers. ESMO Open. 2025 Nov;10(11):105806. doi: 10.1016/j.esmoop.2025.105806. Epub 2025 Oct 23. PMID 41135379
- [Derived] Muro K, Feinstein T, Baranda J, Bonta I, Yanagitani N, Gersten T, Gandhi L, Kudo T, Fujioka N, Kaplan J, Gorla S, Liu S, Wozniak M, Poondru S, Dillon R, Meng C, Patil T. Enfortumab vedotin in patients with advanced non-small cell lung cancer after disease progression on platinum- and PD-1/PD-L1 inhibitor-containing regimens: Phase 2 international multicenter EV-202 study. Eur J Cancer. 2025 Sep 9;227:115603. doi: 10.1016/j.ejca.2025.115603. Epub 2025 Jul 9. PMID 40819431
- [Derived] Swiecicki PL, Yilmaz E, Rosenberg AJ, Fujisawa T, Bruce JY, Meng C, Wozniak M, Zhao Y, Mihm M, Kaplan J, Gorla S, Geiger JL. Phase II Trial of Enfortumab Vedotin in Patients With Previously Treated Advanced Head and Neck Cancer. J Clin Oncol. 2025 Feb 10;43(5):578-588. doi: 10.1200/JCO.24.00646. Epub 2024 Oct 31. PMID 39481054